CLINICAL TRIAL: NCT05343936
Title: Evaluation of an Active Surveillance Protocol for Prostate Cancer in the Brazilian Population
Status: Recruiting | Type: Observational
Sponsor: Hospital Moinhos de Vento (Other)
Responsible Party: Sponsor
Other Study IDs: 56352622.8.1001.5330
Record Dates: First submitted 2022-04-11; First posted 2022-04-25 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
Keywords: active surveillance
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — Paraffin fixed tissue of prostate cancer biopsies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Active surveillance: This is a multicentric active surveillance prospective cohort study. The eligibility criteria defined are: low-risk prostate adenocarcinoma (clinical stage of cT1-T2a / Group Grade 1 (Gleason score less or equal to 6) / PSA less or equal to 10 ng/ml), transrectal prostate biopsy with at least 12 cores, estimated life expectancy over 10 years, clinical conditions for definitive treatment, multiparametric prostate MRI performed or planned.
  Interventions: Other: Active surveillance

INTERVENTIONS:
Other: Active surveillance — The active surveillance protocol involves a TRUS prostate biopsy at eligibility, at 12 months and then every two years. MRI with or without biopsy at eligibility and then every two years. Clinical evaluation with digital rectal examination and PSA every 6 months. Every year a quality of life and anxiety evaluation are planned.
  A new prostate biopsy is indicated if biochemical progression by PSA or changes in multiparametric MRI. Triggers for definitive intervention are biopsy pathological reclassification with Gleason score greater than 6, clinical progression or patient's request.

SUMMARY:
In this study, the investigators aim to form a Brazilian national prospective active surveillance cohort of patients with low-risk prostate cancer in the public health system. The investigators aim to demonstrate data on the pathological reclassification rate, treatment-free survival, among others. This cohort aim to evaluate and validate the active surveillance strategy in Brazil.

DETAILED DESCRIPTION:
Prostate cancer is the most common malignancy in men in Brazil. It is estimated that about 80% of patients diagnosed with prostate cancer have localized disease, and many of these cases have low-risk cancer.

Active surveillance(AS) is a treatment strategy mainly for low risk prostate cancer to avoid radical treatment through periodic assessments (PSA, digital rectal exam and Prostatic Biopsies). During this follow-up, the patient will be treated only when necessary and with curative intent. Several series of institutional cohorts with long-term follow-up have demonstrated that the AS strategy in selected patients is a safe alternative to immediate treatment, with comparable survival.

The active surveillance strategy has never been evaluated in the Brazilian population. The main outcomes from AS derive from international cohorts. The Brazilian population is extremely diverse, so validation in this cohort is relevant. The current study aim to form a national multicentric prospective cohort of patients with low-risk prostate cancer following an AS protocol in the the public health system to evaluate and validate this strategy in Brazil.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of prostate adenocarcinoma;
* Prostate biopsy with at least 12 cores;
* PSA less than or equal to 10 ng/ml and clinical stage cT1/cT2a;
* Gleason score below or equal to 6 (3+3);
* Prostate multi parametric MRI performed or planned
* Availability of pathological samples

Exclusion Criteria:

* Clinical contraindication to prostatectomy and/or radiotherapy procedures;
* Life expectancy below 10 years, according to the Charlson Comorbidity Index (ICC);
* Previous treatment with hormone blockade or radical therapies.
* Intraductal or cribriform histology on biopsy

Ages: 18 Years to 78 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Brazilian men with prostate adenocarcinoma with localized and low-risk disease. They should be attending in the public healthcare system and being treated by the active surveillance protocol.
Sampling Method: Probability Sample
Enrollment: 490 (Estimated)
Dates: Start 2022-08-19 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Biopsy pathological reclassification rate | 12-month analysis
  Gleason score above 6 (min: 6 - max: 10) in prostate biopsy

SECONDARY OUTCOMES:
Treatment-Free Survival rate | 12-month and 24-month analysis
Overall survival rate | 12-month and 24-month analysis
Cancer-Specific Mortality Rate | 12-month and 24-month analysis
Metastasis-free survival rate | 12-month and 24-month analysis
Quality of life evaluation | 12-month and 24-month analysis
  EQ-5D-5L questionnaire
EPIC evaluation | 12-month and 24-month analysis
  Expanded Prostate Cancer Index Composite for Clinical Practice (EPIC-CP) questionnaire (min: 0 - max: 60). Higher scores are worse.
Anxiety evaluation | 12-month and 24-month analysis
  General Anxiety Disorder-7 questionnaire (min: 0 - max: 21) Higher scores are worse
Biochemical recurrence rate after radical therapy | 12-month and 24-month analysis
  PSA greater than or equal to 0.2 ng/ml after radical prostatectomy or PSA nadir plus 2 ng/ml after radiotherapy;

OTHER OUTCOMES:
Monitoring of active surveillance harm | 12-month and 24-month analysis
  Occurrence of any complications in prostate biopsies
Evaluation of pathological outcomes in patients undergoing radical prostatectomy | 12-month and 24-month analysis
  Presence or absence of any of the following criteria: Gleason score above 6 (min: 6 - max: 10), positive surgical margins, extracapsular extension, seminal vesicle invasion or positive lymph node metastases

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Henrique Isaacsson Velho, M.D., Principal Investigator — Head of Clinical Research
Locations (15):
- Brazil (15):
  - Oncocentro Ceará, Fortaleza, Ceará
  - Hospital Universitário Cassiano Antônio Moraes, Vitória, Espírito Santo
  - Hospital Obras de Caridade Irma Dulce, Salvador, Estado de Bahia
  - Hospital Santa Izabel, Salvador, Estado de Bahia
  - Hospital Universitario de Brasilia, Brasília, Federal District
  - Hospital Mario Penna, Belo Horizonte, Minas Gerais
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - Hospital Universitario Joao de Barros Barreto, Belém, Pará
  - Hospital Escola - UFPEL, Pelotas, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceição, Porto Alegre, Rio Grande do Sul
  - Hospital Universidade Dr. Miguel Riet Corrêa Jr., Rio Grande, Rio Grande do Sul
  - Hospital de Amor, Barretos, São Paulo
  - IAMSPE, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Basso J, de Lima JB, Bessel M, Tobar Leitao SA, Machado Baptista T, Roithmann S, Franco Carvalhal E, da Silva Schmitt C, Morzoletto Pedrollo I, Schuch A, Atalibio Hartmann A, Neubarth Estivallet CL, Behrend Silva Ribeiro G, Zordan RA, Isaacsson Velho P. The Brazilian national prospective active surveillance (AS) cohort of patients with low-risk prostate cancer in the public health system: vigiaSUS study protocol. BMC Urol. 2023 Dec 11;23(1):208. doi: 10.1186/s12894-023-01380-w. PMID 38082337